CLINICAL TRIAL: NCT02504021
Title: Family Consultation for High-Risk Inpatients With End Stage Renal Disease: A Randomized Trial
Brief Title: Family Meeting Study for End Stage Renal Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mark A. Lumley (Other)
Collaborators: Henry Ford Health System (Other)
Responsible Party: Sponsor-Investigator, Mark A. Lumley, Professor, Wayne State University
Organization: Wayne State University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HFHS IRB 9714
Record Dates: First submitted 2015-07-14; First posted 2015-07-21 (Estimated); Last update posted 2017-09-19 (Actual); Status verified 2017-09

CONDITIONS: End-stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Family Consultation Condition (Experimental): The family consultation will be one, 1-hour session conducted by trained, master's level therapists. The goals of the meetings are: a) Review patient and family understanding of events that caused the hospital admission; b) increase family awareness of the level of cognitive impairment that the patient is experiencing; c) discuss ways the family can get involved and help the patient with their medication and dialysis adherence; d) use motivational interviewing techniques as needed. This will be provided in addition to the usual care that inpatients receive in this unit.
  Interventions: Behavioral: Family Consultation
- Treatment as Usual Control Condition (No Intervention): Standard of care for the nephrology unit.

INTERVENTIONS:
Behavioral: Family Consultation — This intervention is based on psychoeducation, social support mobilization, and motivational interviewing techniques.
  Arms: Family Consultation Condition

SUMMARY:
A randomized clinical trial for patients with end stage renal disease in which a family consultation condition is compared against a treatment as usual control condition on the hospital readmissions after 1 month as the primary outcome variable.

DETAILED DESCRIPTION:
Patients hospitalized at Henry For Hospital who have end stage renal disease will complete baseline questionnaires and be randomized into the experimental or control condition. Patients randomized into the experimental condition will have a single family consultation session before the patient is discharged. A trained, master's level therapist will conduct the family consultation, which will use education, motivational interviewing, and other techniques to help the family engage and support the patient's health needs. Patients in both the experimental and control conditions will complete follow up questionnaires 1 month after discharge. Investigators will conduct chart reviews of outcome data, including readmissions, at 1, 3, and 6 months post-discharge.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized in inpatient Nephrology Unit at Henry Ford Hospital
* Has end-stage renal disease
* Willing and able to contact support person / family member about participating in the study

Exclusion Criteria:

* Persistent Delirium
* Non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-07; Primary Completion 2016-05 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Early Hospital Readmissions - 1 Month | 1 Month
  Were patients readmitted to the hospital within 1 month of their initial discharge?

SECONDARY OUTCOMES:
Change in Instrumental Social Support | Baseline and 1-month follow-up
  Amount of involvement of support people in terms of disease management. Items modified from the Diabetes Social Support Questionnaire-Family.
Change in Medication Adherence | Baseline and 1-month follow-up
  Adherence to medication regimen. Items modified from Immunosuppressant Therapy Adherence Scale.
Change in Depression | Baseline and 1-month follow-up
  Assessed using Patient Health Questionnaire 8
Change in Anxiety | Baseline and 1-month follow-up
  Assessed using Generalized Anxiety Disorder Questionnaire-7
Change in Biological Measures of Health | Baseline, 1, and 3 months
  Based on chart review, investigators will assess BUN, creatinine, substance use (tox screen), phosphorous, comorbidities, mortality
Hospital Readmissions - 3 Months | 3 Months
  Were patients readmitted to the hospital within 3 months of their initial discharge?

CONTACTS AND LOCATIONS:
Overall Officials: Mark W Ketterer, Ph.D., Principal Investigator — Henry Ford Health Systems
Locations (1):
- Henry Ford Health System, Detroit, Michigan, United States